CLINICAL TRIAL: NCT07023575
Title: Study on Screening Strategies for Interstitial Lung Abnormalities and Airway Lesions
Acronym: SSILA
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Ma Xiao, Chief Physician, China-Japan Friendship Hospital
Other Study IDs: 2024ZD0522301
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Interstitial Lung Abnormalities
Keywords: interstitial lung abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese Routine Chest CT Health Examination Cohort: This group includes individuals who underwent routine health examinations with chest CT imaging at participating health checkup centers across China between 2017 and 2024. Participants may have one or more CT records, and no interventions were applied as part of the study. This group will be analyzed for the presence of interstitial lung abnormalities and/or airway diseases based on imaging and lung function data, as well as demographic and clinical characteristics.

SUMMARY:
The goal of this observational study is to learn about the comorbidity patterns of interstitial and airway abnormalities in adults undergoing health examinations in China. The main questions it aims to answer are:

How do early interstitial lung abnormalities progress to comorbid interstitial and airway diseases? What are the key factors associated with this progression?

Participants undergoing routine health examinations will be assessed for interstitial and airway abnormalities based on imaging and clinical data. Longitudinal follow-up will be used to evaluate disease progression and identify associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Underwent chest CT examination between January 1, 2017 and December 31, 2024
* Age 18 years or older at the time of examination

Exclusion Criteria:

- Missing or incomplete key demographic or imaging information (e.g., missing date of examination, sex, age, or CT report)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from multiple health checkup centers across various regions of China between 2017 and 2024. Specifically, this retrospective study included data from 10 hospital-based health examination institutions located within the four major economic regions of China (East, Central, West, and Northeast). All available health examination records of individuals who underwent chest CT scans during this period were collected for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
high-resolution computed tomography (HRCT) examinations | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongguancun Meinian Health Industry Research Institute, Beijing
  - Central South University, Changsha
  - Affiliated Hospital of Guizhou Medical University, Guiyang
  - Zhejiang University, Hangzhou
  - Henan Provincial People's Hospital, Henan
  - The Affiliated Hospital of Qingdao University, Qingdao
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Henan Hongli Hospital Co., Ltd, Xinxiang

IPD SHARING:
Plan to Share IPD: No